CLINICAL TRIAL: NCT01708486
Title: Multicenter, Prospective, Non-interventional, Observational Study on Treatment of Asthma in Children.
Brief Title: BALLOON (Corticosteroid/laBA inhaLers in adoLescents' Asthma: Assessment Of Patients satisfactiON) Study
Acronym: BALLOON
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-FLUSAL-EL-24
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
Keywords: asthma; Dry Powder Inhalers; FSI-10 questionnaire
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents' with asthma using inhalation devices: Asthmatic adolescents will record their opinion for their inhalation devices by replying to FSI-10 questionnaire

SUMMARY:
Patients' satisfaction with their asthma medication devices is usually decided by using properly designed questionnaires. These questionnaires are to be used to evaluate patients' opinion, which is considered very important for the selection of a device.

The Feeling of Satisfaction with Inhaler (FSI-10) is a self-completed questionnaire designed to assess the patient opinion regarding the satisfaction and usability of the inhalers irrespectively of the drug used. It consists of 10 question each with 5 possible responses on a 5-point Likert scale scored from 5 to 1, respectively. The total score can range between 10 and 50. The higher the score, the higher the feeling of patient satisfaction from the inhaler.

DETAILED DESCRIPTION:
Childhood and adolescents' asthma is the most common chronic disease of childhood and is the major cause of absenteeism from school students. To deal with the disease often require hospitalization, fortunately, very rare enough to be life-threatening. Since the mid-80s had clearly expressed by several centers to observe the rising incidence of the disease. The next year observation was confirmed many times. Childhood asthma has been characterized as a disease of modern Western civilization. It affects a large proportion of the child population and seems to take longer epidemic character.

From studies carried out recently in Greece found that children of school age asthmatic type symptoms during the past 12 months appear to 5-10% of pupils. The rates are doubled when the question is not limited to the last 12 months. Also in a study involving 2133 children aged 7 and 18 years, the prevalence of asthma was 7.7% and 4.7% (at the age of 7 and 18 years respectively) and chronic asthma 19.6% and 26.3% (at the age of 7 and 18 years, respectively), while over half of the children (58.2%) with early asthma (asthma diagnosed before age 7) had no symptoms at the age of 7. At the age of 18 still had symptoms for 7.6% of children with early asthma and 48.2% of children who developed asthma between 7-18 years (6.7% of study participants).

For the onset of childhood asthma synergize two factors: genetic, ie heredity, and environmental, that is the environment in which we live. There is a predisposition for the disease and the environment favors the onset. So to increase the prevalence implicated: a) genetic predisposition, b) the method of construction of houses, c) smoking (assets - liabilities), c) indoor pollution, d) atmospheric pollution, e) the modern way of eating and clothing and f) preventing illness by a large number of serious infections due to the widespread use of vaccines.Most asthma medications are administered using suitable inhalers. There are various types of devices that facilitate the administration of inhaled medications in young children. The correct use of inhalational devices is very important for the treatment of asthma. If the patient does not understand the instructions, the drug is deposited satisfactorily lungs, ie organ must act, so there is no remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of asthma or newly diagnosed
* Patient who are on their inhalation device treatment at least one month before study enrolment
* Patients Male and Female
* Patients' Age: 12-18 years
* Patients who are familiar with their inhalation device
* Patients with correct use of any individual inhalation device
* Patients who will follow all study procedures
* Patients who agree to record their evaluation in written by filling in the FSI-10 questionnaire

Exclusion Criteria:

* Patient who are on their inhalation device treatment less than one month before study enrolment
* Patients' Age: <12, >18 years
* Patients with incorrect use of any individual inhalation device
* Patients with no sufficient treatment compliance
* Patients with no sufficient study procedures' compliance
* Patients who do not agree to record their evaluation in written by filling in the FSI-10 questionnaire

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 180 asthmatic adolescents (60 per device) aged 12-18 years using their inhalation device at least one month before study enrolment. This will be a real-life, regular clinical practice assesment.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feeling of satisfaction with inhalation devices in asthmatic children | 2 months
  FSI-10 questionnaire rating per inhalation device. FSI-10 consists of 10 questions with 5 possible responses on a 5-point Likert scale scored from 5 to 1,respectively. The total score can range between 10 and 50. The higher the score, the higher the feeling of patient satisfaction from the inhaler.

SECONDARY OUTCOMES:
FSI-10 questionnaire ratings' comparison for inhalation devices | 2 months
  The total score will be compared among devices. Each question grating will be also compared among devices.

CONTACTS AND LOCATIONS:
Overall Officials: Ch Hatzimihael, MD Professor, Principal Investigator — Democretion University of Alexandroupolis, Pediatric Department, Thrace, Greece; Emm Paraskakis, MD, Ass Professor, Principal Investigator — Demokretion University of Alexandroupolis, Pediatric Department, Thrace, Greece; Ath Kaditis, MD, Principal Investigator — Agia Sofia Childrens Hospital of Athens, University Pediatric Clinic, Pulmonology Department; Poly Panayotopoulou, MD, Principal Investigator — Agia Sofia Childrens Hospital of Athens, University Pediatric Clinic, Pulmonology Department; Dimos Gidaris, MD Pulmonologist, Principal Investigator — Hippokration Hospital of Thessaloniki, Scientific collaborator; Michael Anthrakopoulos, MD, Associate Professor, Principal Investigator — University Hospital of Rio, Patras, Greece
Locations (1):
- Hippokrateion University Hospital, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Background] Campbell JL, Kiebert GM, Partridge MR. Development of the satisfaction with inhaled asthma treatment questionnaire. Eur Respir J. 2003 Jul;22(1):127-34. doi: 10.1183/09031936.03.00097503. PMID 12882462
- [Background] Kozma CM, Slaton TL, Monz BU, Hodder R, Reese PR. Development and validation of a patient satisfaction and preference questionnaire for inhalation devices. Treat Respir Med. 2005;4(1):41-52. doi: 10.2165/00151829-200504010-00005. PMID 15725049
- [Background] Perpina Tordera M, Viejo JL, Sanchis J, Badia X, Cobos N, Picado C, Sobradillo V, Martinez Gonzalez del Rio J, Duce F, Munoz Cabrera L. [Assessment of patient satisfaction and preferences with inhalers in asthma with the FSI-10 Questionnaire]. Arch Bronconeumol. 2008 Jul;44(7):346-52. Spanish. PMID 18727886
- [Background] Epstein S, Maidenberg A, Hallett D, Khan K, Chapman KR. Patient handling of a dry-powder inhaler in clinical practice. Chest. 2001 Nov;120(5):1480-4. doi: 10.1378/chest.120.5.1480. PMID 11713123
- [Background] van der Palen J, Klein JJ, van Herwaarden CL, Zielhuis GA, Seydel ER. Multiple inhalers confuse asthma patients. Eur Respir J. 1999 Nov;14(5):1034-7. doi: 10.1183/09031936.99.14510349. PMID 10596686
- [Background] Reliability of the FSI-10 questionnaire for the assessment of the usability of drug inhalers in Greek patients. N. Grekas, A. Athanassiou, C. Iskos, D. Panagiotakos, A. Papataxiarchou, O. Porichi. Arch Hellen Med, 28(2), March-April 2011, 257-260.
- See also: Reliability of the FSI-10 questionnaire for the assessmentof the usability of drug inhalers in Greek patients — http://www.mednet.gr/archives/2011-2/pdf/257.pdf